CLINICAL TRIAL: NCT05504785
Title: DexCom Hospital Study-CGM Directed Insulin Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Hip/knee arthroplasty patients are now discharged from hospital within 12 to 24 hours after COVID. patients no longer visited the pre-admission testing center after COVID so unable to insert glucose sensors pre-op.
Sponsor: Thomas Jefferson University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 12039
Record Dates: First submitted 2021-02-25; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes; Hip Osteoarthritis; Knee Osteoarthritis
Keywords: Type 2 diabetes; joint replacement surgery; Insulin dose protocol; Real-time Continuous Glucose Monitor (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Twenty type 2 diabetic patients in the Control Group will be managed according to standard-of-care methods at TJUH using finger-stick blood glucose measurements in an attempt to maintain the patient's blood glucose levels in the desired target range (80 to 180 mg/dL).
  Forty type 2 diabetic patients in the Investigational Group will be managed by the orthopedic floor nurses using the real-time DexCom G6 CGM trend data and an insulin dosing protocol to determine the appropriate therapy to maintain the patient's glucose levels in the desired target range (80 to 180 mg/dL). T
  Glucose control will be compared between the two groups, and glucose control will be correlated with post-operative clinical adverse events (wound infection, deep vein thrombosis, pulmonary embolism, extended hospital LOS, hospital re-admission, emergency room visit).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group (Active Comparator): Twenty type 2 diabetic patients in the Control Group will be managed according to standard-of-care methods at TJUH using finger-stick blood glucose measurements in an attempt to maintain the patient's blood glucose levels in the desired target range (80 to 180 mg/dL). Three blinded CGM will be used to record the patient's glucose trend data (for 20 days maximum) for future download to a computer and analysis.
  Interventions: Device: DexCom G6 continuous glucose monitor
- Investigational Group (Active Comparator): Forty type 2 diabetic patients in the Investigational Group will be managed by the orthopedic floor nurses using the real-time DexCom G6 CGM trend data to determine the appropriate therapy to maintain the patient's glucose levels in the desired target range (80 to 180 mg/dL). In addition, three blinded CGM will be used to record the patient's glucose trend data (for 20 days maximum) for future download to a computer and analysis.
  Interventions: Device: DexCom G6 continuous glucose monitor

INTERVENTIONS:
Device: DexCom G6 continuous glucose monitor — Use of real-time DexCom G6 continuous glucose monitor (CGM or glucose sensor) trend data and an insulin-dosing algorithm to control the glucose levels of diabetic patients undergoing hip/knee orthopedic surgery at Thomas Jefferson University Hospital (TJUH).

SUMMARY:
This is a pilot investigator initiated/sponsored clinical trial to evaluate the feasibility of using real-time DexCom G6 continuous glucose monitor (CGM or glucose sensor) trend data and an insulin-dosing algorithm to control the glucose levels of type 2 diabetic patients undergoing hip/knee orthopedic surgery at Thomas Jefferson University Hospital (TJUH).

Blinded CGM glucose data will be recorded prior to hospital admission, during hospital admission, and after hospital discharge to evaluate glucose control in this diabetic patient population in relationship to clinical outcomes (20 days of recorded blinded CGM data maximum). Prior studies have associated hyperglycemia, hypoglycemia, and glycemic variability with an increased incidence of nosocomial infection, deep vein thrombosis, pulmonary embolism, cardiac arrhythmias, mental status changes, hospital length of stay, and cost.

The 20 type 2 diabetic patients in the Control Group will be managed according to standard-of-care methods at TJUH using finger-stick blood glucose measurements in an attempt to maintain the patient's blood glucose levels in the desired target range (80 to 180 mg/dL). Three blinded CGM will be used to record the patient's glucose trend data for future download to a computer and analysis.

The 40 type 2 diabetic patients in the Investigational Group will be managed by the orthopedic floor nurses using the real-time DexCom G6 CGM trend data to determine the appropriate therapy to maintain the patient's glucose levels in the desired target range (80 to 180 mg/dL). In addition, three blinded CGM will be used to record the patient's glucose trend data for future download to a computer and analysis.

The primary objective of this pilot study is to observe the blood glucose values and glucose sensor (CGM) values of diabetic patients before, during and after hospitalization for hip and knee arthroplasty surgery to determine whether there is a correlation between glucose control and clinical outcomes. This pilot data will be used to plan a future clinical trial in orthopedic surgery patients using CGM to determine patterns of hyperglycemia, hypoglycemia, and glycemic variability that correlate with clinical complications, hospital length of stay, and cost.

DETAILED DESCRIPTION:
The investigators hypothesize that real-time CGM trend data can be used by the hospital floor nurse to safely dose insulin to maintain the glucose concentration in the target range (80-180 mg/dl), minimize the risk for mild hypoglycemia (< 70 mg/dL), and eliminate the risk for severe hypoglycemia (<54 mg/dL).

Subjects may be consented during their pre-operative visit to the TJUH Pre-Admissions Testing Center (PAT) or during their pre-operative visit to the Department of Orthopedic Surgery's outpatient Rothman Clinic. Twenty patients with type 2 diabetes will be assigned to a control group (n=20) and forty patients will be assigned to an investigational group (n=40).

The skin surface around each CGM insertion site may be photographed; then prepped with alcohol/chlorhexidine and allowed to dry. Research personnel will insert 3 blinded Dexcom G6 CGM into the upper arm (n=1) and abdomen/flank (n=2) of each study subject using sterile gloves and aseptic technique. The 3 blinded CGM will measure and record the concentration of tissue fluid glucose every 5 minutes for up to 10 days.

Control Group (Hospital Admission):

Blinded CGM that were inserted more than 8 or 9 days ago will be removed by research personnel prior to surgery Three new blinded DexCom G6 CGM will be inserted into an alternate location of the study subject's upper arm (n=1) and abdomen/flank (n=2) using aseptic technique.

Patients may be discharged from the hospital approximately 24 to 48 hours after the surgical procedure wearing 3 blinded CGM. Patients will be instructed to self-remove the 3 blinded CGM after a maximum of 10 days of wear-time, and place the blinded CGM into a plastic specimen cup and a stamped addressed envelope. Subjects will be instructed to mail the envelop to TJU research personnel.

Investigational Group (Hospital Admission):

Blinded CGM that were inserted more than 8 or 9 days ago will be removed by research personnel prior to surgery in the SDA Uni. Two new blinded DexCom G6 CGM will be inserted into an alternate location of the study subject's upper arm (n=1) and abdomen/flank (n=2) using aseptic technique. One new real-time Dexcom G6 CGM will be inserted into the subcutaneous tissue of the abdomen using aseptic technique The real-time CGM will be activated and coupled to a tablet computer for data display at the bedside. The iPad will be programmed to alarm if the CGM glucose falls below < 90 mg/dL (threshold alarm) or if the CGM predicts the glucose concentration will fall below < 55 mg/dL in the next 20 minutes (predictive alarm).

Patients may be discharged from the hospital approximately 24 to 48 hours after the surgical procedure wearing 3 blinded CGM. They will be instructed to self-remove the 3 blinded CGM after a maximum of 10 days of wear-time, and place the blinded CGM in a plastic cup and stamped addressed envelope. Subjects will be instructed to mail the envelope to TJU research personnel.

In-hospital Glucose Control Methods (Control Group):

The control group of patients will be managed using routine standard-of-care TJUH methods. Study subjects will have fingerstick blood glucose (BG) measurements performed before breakfast, before lunch, before dinner, at 9:00pm and 2:00am (5 assessments per day) using a commercial meter and test strips. The floor nurse may obtain additional finger stick BG measurements at any time to detect or confirm hypoglycemia/hyperglycemia. Diabetic patients will be managed by their orthopedic surgeons (with input from the endocrinologists) using the oral anti-diabetic medications and/or long-acting and rapid-acting insulin injections routinely used at home.

In-hospital Glucose Control Methods (Investigational Group):

The blood glucose management of the investigational group of diabetic patients will be per the usual practice of the Thomas Jefferson University Hospital (TJUH) orthopedic surgeons. Some of the investigational study subjects will be managed with oral anti-diabetic medications as their baseline diabetes therapy in the hospital, while other subjects will be managed with intermittent injections of long-acting insulin and/or rapid acting insulin with meals. This baseline diabetes therapy will be adjusted based upon the standard-of-care TJUH Correction Dose Insulin Therapy protocol.

The orthopedic floor nurses will make an assessment using the real-time CGM trend data before each meal and 2-hours after each meal. More or less correction dose insulin will be injected into the patient's subcutaneous tissue, based upon the real-time CGM glucose measurement (mg/dL), direction of change, and rate of change. An additional nursing assessment will be made at 9 pm and 2 am using the real-time CGM glucose measurement to determine if the glucose concentration is greater than 300 mg/dL.

The orthopedic nurses will use the displayed real-time CGM trend data (absolute glucose measurement, direction of change, and rate of change) to modify the correction dose of rapid acting insulin according to the TJUH Correction Dose Insulin (CDI) Protocol. The orthopedic floor nurse will assess the real-time displayed CGM trend data before breakfast, 2-hours after breakfast, before lunch, 2-hours after lunch, before dinner, 2-hours after dinner, at 9:00 pm and at 2:00 am (8 nursing assessments per day).

Pre-meal Assessment:

The orthopedic surgery floor nurse will make an assessment using the real-time CGM absolute glucose value (mg/dL) and the CGM direction/rate-of-change glucose trend data (↑-↓ arrows) prior to each meal to determine the correction dose of rapid acting insulin. The correction dose of rapid acting insulin (lispro) will be added or subtracted from the dose of insulin routinely ordered by the orthopedic surgeon to cover the meal. Several examples of pre-meal assessments and insulin dose calculations are provided below.

Post-meal Assessments:

The orthopedic floor nurse will utilize the displayed real-time CGM trend data to determine the correction dose of insulin to be injected 2-hours after each meal. (2-hours after the pre-meal insulin injection). This additional correction insulin dose of insulin may be given two hours after the meal if the GCM data displays hyperglycemia (CGM > 150 mg/dL) with an increasing rate of change. Several examples of post-meal assessments and insulin dose calculations are provided below. An additional correction insulin dose of insulin may be given at 9 pm and/or 2 am only if the CGM displays a glucose concentration > 300 mg/dL.

CGM Alarms For Hypoglycemia:

The orthopedic floor nurse will have the study subject consume 15 grams of oral glucose (tablets or gel) if the real-time CGM alarms for predicted hypoglycemia (CGM < 55 mg/dl predicted 20 minutes in the future) or hypoglycemia below a threshold value (CGM < 80 mg/dL). The orthopedic nurse will make an assessment using the real-time CGM data display approximately 15-20 minutes after the hypoglycemia treatment to confirm the CGM glucose measurements remains > 80 mg/dL. An addition 15 grams of oral glucose will be given approximately 15-20 minutes after the initial oral glucose treatment if the CGM measurement does not remain > 80 mg/dL. If unable to consume oral glucose or altered consciousness, the nurse will treat the hypoglycemia with an intravenous injection of 25 ml dextrose 50% (12.5 grams) or 1 mg glucagon IM/SC based upon the standard-of-care methods used at TJUH to treat hypoglycemia (Table # 3).

Finger Stick BG Measurements:

Study subjects in the Investigational Group will have finger stick capillary blood glucose (BG) measurements performed using a hospital meter/test strips before breakfast, before lunch, before dinner, at 9:00pm, and at 2:00am (5 per day). The nurse may obtain additional finger stick BG measurements at any time to detect or confirm accuracy of the CGM measure and to confirm hypoglycemia/hyperglycemia. All finger stick BG measurement will be recorded in the electronic medical record (EPIC).

Hospital Discharge:

Study subjects will wear the 3 blinded CGM at home during their daily activities for a maximum of 10 days (from date of insertion). Subjects will be instructed to self-remove the blinded 3 CGM after a maximum of 10 days of wear-time, and place the blinded CGM in a stamped addressed envelope. Subjects will be instructed to mail the addressed envelope to TJU research personnel. Research Personnel will contact each study subject by telephone after CGM removal to confirm no serious device related adverse events.

Orthopedic Surgery Medical Record Review:

The hospital and orthopedic surgeon's medical record of each patient will be evaluated following the post-operative visit at the Department of Orthopedic Surgery's Rothman Institute. The medical record review will determine whether there were any adverse events or complications related to the hip/knee surgical procedure (surgical site infection, urinary tract infection, lower respiratory tract infection, myocardial infarction, deep vein thrombosis, pulmonary embolism, stroke, kidney failure, death, emergency room visit, and hospital re-admission).

ELIGIBILITY:
Inclusion Criteria:

* All type 2 diabetic patients undergoing a single surgical hip or knee replacement at Thomas Jefferson University Hospital (TJUH); on an outpatient regimen of oral antidiabetic medication, injectable antidiabetic medication, basal-bolus insulin therapy, or premix insulin therapy.
* Age 30 to 80 years
* BMI ≤ 40

Exclusion Criteria:

* BMI > 40.
* Age < 30 years or > 80 years
* History of two of more hypoglycemia episodes in last 12 months.
* History of severe hypoglycemia unawareness.
* History of diabetic ketoacidosis (DKA) in the last 6 months.
* History of significant skin/tissue reaction (irritation or allergy) to the Continuous Glucose Monitor's (CGM) adhesive tape, plastic bandage, or chlorhexidine.
* Skin infection or disease at the site of CGM insertion.
* Moderate or severe systemic immune deficiency (previous 90 days).
* Currently enrolled in any industry sponsored medical device or pharmaceutical research clinical trial.
* Treated with high-dose anticoagulation therapy at the time of CGM insertion.
* Double or revision knee/hip replacement surgery.
* Anticipate an MRI is required during the hospitalization.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Observe correlation of glucose control and post-operative adverse clinical events | perioperative period x 60 days
  Observe blood glucose values and continuous glucose monitor (CGM or glucose sensor) values of diabetic patients before, during and after hospitalization for joint arthroplasty surgery to determine whether there is a correlation between glucose control and clinical outcomes. CGM data (mg/dL, mean, median, standard deviation, percent of 24 hours within the target range (80-180 mg/dL), above the target range (180-240 mg/dL and > 240 mg/dL), and below the target range (< 70 mg/dL, 40-70 mg/dL, < 40 mg/dL) will be correlated with the incidence of wound infection, deep vein thrombosis, pulmonary embolism, extended hospital length of stay, hospital re-admission, and post-op emergency room visits. Finger-stick blood glucose measurements will also be correlated with adverse clinical outcomes.

SECONDARY OUTCOMES:
Hospital nurses and physicians provide subjective feedback regarding the ease-of-use and human-factors issues following clinical use of the real-time CGM trend data | perioperative period x 1 to 3 days
  Real-time CGM trend data will be used by the post-operative floor nurses to determine/calculate each correction dose of insulin (CDI) to improve glucose control and eliminate severe hypoglycemia.
  Nurses and physicians will complete a questionnaire with yes/no questions related to human factors, ease-of use, and integration into the working environment after using the real-time glucose sensor trend data to calculate insulin doses.
Compare the CGM and Accu-Chek time-match glucose measurements | perioperative x 1 to 3 days
  Compare the simultaneous three CGM glucose measurements to each other and to the fingerstick BG measurements made using a hospital Accu-Chek Inform meter and test strips.
  Time-matched CGM glucose measurements will be compared to finger-stick BG measurements using mean absolute relative difference (MARD), Bland-Altman bias plots, and traditional error grid analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Joseph, DO, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No